CLINICAL TRIAL: NCT01068041
Title: Effects of PH3 in Diabetic Nephropathy
Acronym: PH3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PhytoHealth Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PH-CP016
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Placebo Comparator): Placebo
  Interventions: Drug: PH3
- B (Active Comparator): 250mg active ingredient
  Interventions: Drug: PH3
- C (Active Comparator): 500mg active ingredient
  Interventions: Drug: PH3
- D (Active Comparator): 1000mg active ingredient
  Interventions: Drug: PH3

INTERVENTIONS:
Drug: PH3 — Each PH3 tablet, 530 mg/tablet, contains 250 mg of active ingredient. The placebo tablet contains no active ingredient.

SUMMARY:
The primary objective of this clinical study is to evaluate the effectiveness and safety of PH3 for patients with diabetic nephropathy.

The secondary objectives are to identify the optimal dosage for subsequent studies and to provide basis for the next confirmatory study in study design, endpoints, and study methodologies.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females between 18 and 70 years of age with type 1 or type 2 diabetes
2. Sitting blood pressure of <=140/90 mm Hg
3. Serum creatinine <=2.0 mg/dL
4. Urinary albumin: creatinine ratio between 30 mg/g to 1000 mg/g creatinine (of the first urine sample of the day)
5. Hemoglobin A1c <=8%
6. Women of child-bearing potential must test negative in a pregnancy test and take contraception measures to prevent pregnancy and can not be breast-feeding
7. Voluntary written consent to participate in this study

Exclusion Criteria:

1. History of major cardiovascular or cerebrovascular events within 6 months prior to screening
2. History of cancer
3. Receiving chronic nonsteroidal anti-inflammatory therapy
4. History of diabetic ketoacidosis
5. Has clinically significant deviation from normal physical examination findings that, in the principal investigator's judgment, may interfere with the study evaluation or affect subject safety
6. Has participated in other investigational trials within 28 days prior to study enrollment
7. Has taken herbal medical treatment as prescription medication and/or over-the- counter medication, within 28 days prior to study enrollment.
8. Has known allergy to the study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-08; Primary Completion 2014-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Urinary Albumin/Creatinine Ratio (UACR) | 24 weeks

SECONDARY OUTCOMES:
Urine Albumin Serum Creatinine and the estimated GFR (glomerular filtration rate) HbA1c | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wu Chang Yang, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Yi-Jen Hung, MD, Principal Investigator — Tri-Service General Hospital; Huey-Herng Sheu, MD, PhD, Principal Investigator — Taichung Veterans General Hospital
Locations (3):
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei